CLINICAL TRIAL: NCT05213052
Title: Document Magnitude and Timing for Pain Relief of Topical Cream
Brief Title: Effects of Topical Cream for Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 173-001
Record Dates: First submitted 2021-08-31; First posted 2022-01-28 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Floderm topical cream

STUDY DESIGN:
Intervention Model Description: An open-label study design where all study participants will receive the active test product and no placebo is used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Topical cream, 1 - 2 times daily (Experimental): Application of a pea-sized amount of cream applied to skin over the area with chronic pain
  Interventions: Other: Topical cream

INTERVENTIONS:
Other: Topical cream — Topical cream applied to painful joint or muscle

SUMMARY:
To perform a clinical proof-of-concept study on a novel topical formula for pain relief.

DETAILED DESCRIPTION:
An open-label study where each participant will be involved in the study for 4 weeks. During the study participants will use the topical cream 1-2 times daily on the anatomical area(s) causing the most pain.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 34.9 kg/m2 (inclusive)
* Chronic joint/muscle related pain for at least past 6 months
* Experiencing chronic pain in at least one specific anatomical area for more than 6 months.

Exclusion Criteria:

* Cancer during past 12 months
* Chemotherapy during past 12 months
* Currently taking prescription pain medications
* Getting regular joint injections (such as cortisone shots);
* Immunization during last month
* Participation in another clinical trial study during this trial, involving an investigational product or lifestyle change
* Regularly experiencing headaches, including migraines
* Serious active illness within past 6 months
* Significant active uncontrolled illness (such as lymphoma, liver disease, kidney failure, heart failure).
* Skin allergies related to ingredients in test product.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in degree of pain | 4 weeks
  Pain questionnaire - yes/no, score 0-24 hours

SECONDARY OUTCOMES:
Activity level | 4 weeks
  Activities of daily living questionnaire

OTHER OUTCOMES:
Wellness | 4 weeks
  Wellness questionnaire - Score 0-10 [0 being strongly disagree, 10 being strongly agree]

CONTACTS AND LOCATIONS:
Locations (1):
- Gitte Jensen, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No